CLINICAL TRIAL: NCT05830942
Title: Cognitively Engaging Walking Exercise and Neuromodulation to Enhance Brain Function in Older Adults
Brief Title: Up-2 Study: Cognitively Engaging Walking Exercise and Neuromodulation to Enhance Brain Function in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202300001; PRO00046897 (Other: UFIRST); R01AG081477 (NIH); 1R01AG081477-01 (NIH); IRB202300002 (Other: University of Florida IRB)
Record Dates: First submitted 2023-04-11; First posted 2023-04-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Dysfunction; Mobility Limitation; Frail Elderly
MeSH Terms: conditions — Cognitive Dysfunction; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Walking Exercise plus active tDCS (Active Comparator): The walking exercise will focus on use of complex walking tasks such as obstacle crossing, accurate foot placement, and walking on compliant surfaces. Each session will consist of 30 minutes of walking. Active tDCS will be delivered over prefrontal cortex.
  Interventions: Behavioral: Walking Exercise; Device: Prefrontal Active tDCS
- Walking Exercise plus sham tDCS (Sham Comparator): The walking exercise will focus on use of complex walking tasks such as obstacle crossing, accurate foot placement, and walking on compliant surfaces. Each session will consist of 30 minutes of walking. Sham tDCS will be delivered over prefrontal cortex.
  Interventions: Behavioral: Walking Exercise; Device: Prefrontal Sham tDCS

INTERVENTIONS:
Behavioral: Walking Exercise — aerobic walking exercise using complex (cognitively engaging) walking tasks
Device: Prefrontal Active tDCS — 20 minutes of 2 milliamp transcranial direct current stimulation (tDCS) of prefrontal regions, delivered at each session
  Arms: Walking Exercise plus active tDCS
Device: Prefrontal Sham tDCS — 30 seconds of 2 milliamp transcranial direct current stimulation (tDCS) of prefrontal regions, delivered at each session
  Arms: Walking Exercise plus sham tDCS

SUMMARY:
Declines in cognitive function and walking function are highly intertwined in older adults. A therapeutic approach that combines complex (cognitively engaging) aerobic walking exercise with non-invasive electrical brain stimulation may be effective at restoring lost function. This study tests whether electrical stimulation of prefrontal brain regions is more beneficial than sham stimulation.

DETAILED DESCRIPTION:
Efficacy of transcranial direct current stimulation (tDCS) combined with complex (cognitively engaging) walking exercise in older adults. The primary outcome measures are executive function (computer-based assessment battery) and complex walking function (speed on an obstacle negotiation task). This will be a two-site trial conducted at the University of Florida (lead site) and Brooks Rehabilitation Hospital, which is necessary to achieve enrollment targets and will allow us to develop a multi-site research infrastructure for a future Phase 3 multi-site trial. The study will enroll up to 120 older adult women and men, who exhibit mild to moderate decline of executive function. All experimental groups will receive the same complex walking intervention, which will focus on use of cognitively engaging tasks such as obstacle crossing, accurate foot placement, and walking on complaint surfaces. Each session will consist of 30 minutes of walking. For tDCS, the active treatment group will receive 20 minutes of 2mA tDCS over prefrontal regions F3/F4 ("treatment group"). The second group is a sham control group. tDCS will be delivered simultaneously with complex walking exercise for 18 sessions over a 6-week period. Assessments will be conducted at baseline, post intervention (within one week), and 12 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Objective executive function decline, based on standardized cognitive assessments.
* Subjective cognitive decline, based on the question: "During the past 12 months, have you experienced confusion or memory loss that is happening more often or getting worse?"
* Ability to walking independently for 6 minutes (use of cane permitted)

Exclusion Criteria:

* Major cognitive disorder that interferes with independence
* Percentile score less than 10th percentile on standardized cognitive assessments
* Medications that are thought to influence tDCS neuroplasticity.
* Contraindications to tDCS or MRI.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
walking speed for obstacle task negotiation task | baseline, post-intervention (an average of 6 weeks after baseline), follow-up (an average of 12 weeks after post-intervention)
  change in walking speed from baseline to post intervention (or follow-up) timepoint
score on test of executive function | baseline, post-intervention (an average of 6 weeks after baseline), follow-up (an average of 12 weeks after post-intervention)
  change in score from baseline to post intervention (or follow-up) timepoint

CONTACTS AND LOCATIONS:
Overall Officials: David J Clark, ScD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Brooks Rehabilitation, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No